CLINICAL TRIAL: NCT03821818
Title: Food Allergen Eliminations and Combined Protocols for Obesity Reduction: a Preliminary Comparison Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Galveston Clinical Research Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: 2018.04
Record Dates: First submitted 2018-05-31; First posted 2019-01-30 (Actual); Last update posted 2019-01-30 (Actual); Status verified 2019-01

CONDITIONS: Obesity
Keywords: Food Hypersensitivity; Exercise
MeSH Terms: conditions — Obesity; Food Hypersensitivity; Motor Activity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control: Food Allergen Elimination only
- Allergen Elimination + Willis Exercise: Subjects will have food allergens eliminated and also perform Aerobic-surge, brief high intensity exercise > 75% max HR), five times/day.
  Interventions: Behavioral: Food Allergy Elimination + Willis Exercise

INTERVENTIONS:
Behavioral: Food Allergy Elimination + Willis Exercise — Food Allergy Elimination + Willis Exercise (performing a 2-minute Aerobic-surge exercise > 75% max heart rate, 5/day)
  Other Names: Willis exercise
  Groups: Allergen Elimination + Willis Exercise

SUMMARY:
Screened subjects will be tested for hidden food allergies. Subjects will eliminate all food that showed leukocyte reactions for 90-days. Subjects will then also be invited to use the Willis Exercise protocol. Body composition testing and Body Mass Index calculation will be accomplished at enrollment and after completion of the 90-day study.

DETAILED DESCRIPTION:
Subjects will first be screened for cardiovascular pathologies and then tested for hidden food allergies. After the results subjects will eliminate all food that showed leukocyte reactions for 90-days. Subjects will then also be invited to use the Willis Exercise protocol (Aerobic-surge exercise > 75% max heart rate, for 2-minutes, 5/day. Body composition testing and Body Mass Index calculation will be accomplished at enrollment and after completion of the 90-day study.

ELIGIBILITY:
Inclusion Criteria:

1. The subject is > 20 years of age and is willing and able to provide signed informed consent.
2. The subject has a BMI > 30.
3. The subject is between the ages of 20 to 75 years of age.

Exclusion Criteria:

1. Cardiovascular Heart Disease and this includes but is not limited to history of myocardial infarction, atrial fibrillation, etc.
2. History of cerebral vascular event (stroke), traumatic brain injury, Parkinson's disease or any other neural injury or disease.
3. Diabetes Mellitus (Type I or II)
4. Pregnancy
5. Participation in any other weight loss protocols, diets, or medication.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy, obese subjects
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2018-03-05 (Actual); Primary Completion 2018-08-15 (Actual); Study Completion 2019-08-30 (Estimated)

PRIMARY OUTCOMES:
Change in Body Weight | 90-days
  measure Kg

SECONDARY OUTCOMES:
Change in Body Fat % | 90-days
  Percentage of fat vs lean mass
Change in Body Mass Index (BMI) | 90-days
  BMI calculation

CONTACTS AND LOCATIONS:
Overall Officials: Frank B Willis, MBBS, PhD, Principal Investigator — Galveston Clinical Research Foundation
Locations (1):
- Galveston Clinical Research Foundation, Galveston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alpay K, Ertas M, Orhan EK, Ustay DK, Lieners C, Baykan B. Diet restriction in migraine, based on IgG against foods: a clinical double-blind, randomised, cross-over trial. Cephalalgia. 2010 Jul;30(7):829-37. doi: 10.1177/0333102410361404. Epub 2010 Mar 10. PMID 20647174
- [Background] Aydinlar EI, Dikmen PY, Tiftikci A, Saruc M, Aksu M, Gunsoy HG, Tozun N. IgG-based elimination diet in migraine plus irritable bowel syndrome. Headache. 2013 Mar;53(3):514-25. doi: 10.1111/j.1526-4610.2012.02296.x. Epub 2012 Dec 6. PMID 23216231
- [Background] Kesman RL, Ebbert JO, Harris KI, Schroeder DR. Portion control for the treatment of obesity in the primary care setting. BMC Res Notes. 2011 Sep 9;4:346. doi: 10.1186/1756-0500-4-346. PMID 21906302
- [Background] Torbahn G, Gellhaus I, Koch B, von Kries R, Obermeier V, Holl RW, Fink K, van Egmond-Frohlich A. Reduction of Portion Size and Eating Rate Is Associated with BMI-SDS Reduction in Overweight and Obese Children and Adolescents: Results on Eating and Nutrition Behaviour from the Observational KgAS Study. Obes Facts. 2017;10(5):503-516. doi: 10.1159/000480517. Epub 2017 Oct 31. PMID 29084405
- [Background] Iwao S, Mori K, Sato Y. Effects of meal frequency on body composition during weight control in boxers. Scand J Med Sci Sports. 1996 Oct;6(5):265-72. doi: 10.1111/j.1600-0838.1996.tb00469.x. PMID 8960647
- [Background] Fisher G, Brown AW, Bohan Brown MM, Alcorn A, Noles C, Winwood L, Resuehr H, George B, Jeansonne MM, Allison DB. High Intensity Interval- vs Moderate Intensity- Training for Improving Cardiometabolic Health in Overweight or Obese Males: A Randomized Controlled Trial. PLoS One. 2015 Oct 21;10(10):e0138853. doi: 10.1371/journal.pone.0138853. eCollection 2015. PMID 26489022
- [Background] Harris NK, Dulson DK, Logan GRM, Warbrick IB, Merien FLR, Lubans DR. Acute Responses to Resistance and High-Intensity Interval Training in Early Adolescents. J Strength Cond Res. 2017 May;31(5):1177-1186. doi: 10.1519/JSC.0000000000001590. PMID 27537411
- [Background] Irwin ML, Yasui Y, Ulrich CM, Bowen D, Rudolph RE, Schwartz RS, Yukawa M, Aiello E, Potter JD, McTiernan A. Effect of exercise on total and intra-abdominal body fat in postmenopausal women: a randomized controlled trial. JAMA. 2003 Jan 15;289(3):323-30. doi: 10.1001/jama.289.3.323. PMID 12525233
- [Background] Jakicic JM, Otto AD. Treatment and prevention of obesity: what is the role of exercise? Nutr Rev. 2006 Feb;64(2 Pt 2):S57-61. doi: 10.1111/j.1753-4887.2006.tb00235.x. PMID 16532900
- [Background] Sijie T, Hainai Y, Fengying Y, Jianxiong W. High intensity interval exercise training in overweight young women. J Sports Med Phys Fitness. 2012 Jun;52(3):255-62. PMID 22648463
- [Background] Stoner L, Rowlands D, Morrison A, Credeur D, Hamlin M, Gaffney K, Lambrick D, Matheson A. Efficacy of Exercise Intervention for Weight Loss in Overweight and Obese Adolescents: Meta-Analysis and Implications. Sports Med. 2016 Nov;46(11):1737-1751. doi: 10.1007/s40279-016-0537-6. PMID 27139723
- [Background] Warburton DE, Nicol CW, Bredin SS. Health benefits of physical activity: the evidence. CMAJ. 2006 Mar 14;174(6):801-9. doi: 10.1503/cmaj.051351. PMID 16534088
- [Background] Willis FB, Smith FM, Willis AP. Frequency of exercise for body fat loss: a controlled, cohort study. J Strength Cond Res. 2009 Nov;23(8):2377-80. doi: 10.1519/JSC.0b013e3181b8d4e8. PMID 19826285
- [Background] Poulsen SK, Due A, Jordy AB, Kiens B, Stark KD, Stender S, Holst C, Astrup A, Larsen TM. Health effect of the New Nordic Diet in adults with increased waist circumference: a 6-mo randomized controlled trial. Am J Clin Nutr. 2014 Jan;99(1):35-45. doi: 10.3945/ajcn.113.069393. Epub 2013 Nov 20. PMID 24257725
- [Background] Palmer DJ, Huang RC, Craig JM, Prescott SL. Nutritional influences on epigenetic programming: asthma, allergy, and obesity. Immunol Allergy Clin North Am. 2014 Nov;34(4):825-37. doi: 10.1016/j.iac.2014.07.003. Epub 2014 Aug 21. PMID 25282294
- [Background] Hurtado-Barroso S, Tresserra-Rimbau A, Vallverdu-Queralt A, Lamuela-Raventos RM. Organic food and the impact on human health. Crit Rev Food Sci Nutr. 2019;59(4):704-714. doi: 10.1080/10408398.2017.1394815. Epub 2017 Nov 30. PMID 29190113
- [Background] Pergola G, Foroni F, Mengotti P, Argiris G, Rumiati RI. A neural signature of food semantics is associated with body-mass index. Biol Psychol. 2017 Oct;129:282-292. doi: 10.1016/j.biopsycho.2017.09.001. Epub 2017 Sep 9. PMID 28899747

DOCUMENTS (1):
  • Study Protocol (2018-02-01): https://cdn.clinicaltrials.gov/large-docs/18/NCT03821818/Prot_000.pdf